CLINICAL TRIAL: NCT03464344
Title: COrtical Superficial Siderosis and REcurrent Lobar Intracerebral Hemorrhage in Cerebral Amyloid Angiopathy.
Brief Title: Cortical Superficial Siderosis and Risk of Recurrent Intracerebral Hemorrhage in Cerebral Amyloid Angiopathy.
Acronym: CORELIA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: RC31/16/8919; 2017-A01524-49 (Other: ID-RCB)
Record Dates: First submitted 2018-03-07; First posted 2018-03-14 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Cerebral Amyloid Angiopathy
Keywords: intracerebral hemorrhage; cerebral amyloid angiopathy; cortical superficial siderosis; Magnetic Resonance Imaging
MeSH Terms: conditions — Cerebral Amyloid Angiopathy; Cerebral Hemorrhage

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients with cortical superficial siderosis. (Other): During a systematic follow-up of 24 months, patients will undergo neurological, neuropsychological and MRI evaluation
  Interventions: Other: neurological, neuropsychological and MRI evaluation
- Patients without cortical superficial siderosis (Other): During a systematic follow-up of 24 months, patients will undergo neurological, neuropsychological and MRI evaluation
  Interventions: Other: neurological, neuropsychological and MRI evaluation

INTERVENTIONS:
Other: neurological, neuropsychological and MRI evaluation — neurological, neuropsychological and MRI evaluation

SUMMARY:
Cerebral amyloid angiopathy (CAA) is a major cause of lobar intracerebral hemorrhage (ICH) in the elderly with high risk of recurrence.

The investigators aim to determine the relationship between cortical superficial siderosis (cSS), a MRI hemorrhagic marker of CAA and the risk of symptomatic ICH recurrence in a multicentric prospective cohort of patients with acute lobar ICH related to CAA. The investigators hypothesize that patients with cSS have an increased risk of recurrent symptomatic ICH relative to those without cSS.

DETAILED DESCRIPTION:
Patients with acute lobar ICH fulfilling the Boston criteria for probable or possible CAA will be enrolled within 30 days after ICH onset. Brain MRI performed at baseline will be analyzed blinded to clinical data. Patients with presence of cSS will be compared with those without cSS.

During a systematic follow-up of 24 months, patients will undergo neurological, neuropsychological and MRI evaluation. The investigators will compare the rate of recurrent symptomatic ICH at 24 months in patients with vs. without cSS.

ELIGIBILITY:
Inclusion Criteria:

* Lobar ICH within 30 days after onset
* Available brain MRI sequences of adequate quality including fluid-attenuated inversion recovery (FLAIR) and T2*-weighted gradient-recalled echo (T2*-GRE) sequences.
* Modified Boston criteria for probable or possible CAA
* Age ≥ 55 years
* Written consent

Exclusion Criteria:

* Secondary brain hemorrhage : vascular malformation (arteriovenous malformation, aneurysm, cavernous); cerebral veinous thrombosis; brain tumor; coagulopathy; vasculitis; hemorrhagic infarction,
* Infratentorial siderosis
* Contraindications to MRI
* Neurosurgical intervention before inclusion,
* Progressive neoplasm
* Patient without affiliation to the french social security
* Patient under guardianship

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Actual)
Dates: Start 2018-10-12 (Actual); Primary Completion 2025-02-11 (Actual); Study Completion 2025-02-11 (Actual)

PRIMARY OUTCOMES:
Recurrent symptomatic intracerebral hemorrhage at 24 months | 24 months
  Recurrent symptomatic intracerebral haemorrhage is defined as a further intracerebral hemorrhage documented by CT scan or MRI, associated with new neurologic symptoms

SECONDARY OUTCOMES:
Recurrent symptomatic ICH at 12 months | 12 months
  Recurrent symptomatic intracerebral haemorrhage is defined as a further intracerebral hemorrhage documented by CT scan or MRI, associated with new neurologic symptoms.
Transient Focal Neurological Episodes (TFNE) at 12 and 24 months | 12 and 24 months
  TFNE was defined as transient (≤24 hours), with fully resolving, focal neurological symptoms that had no known alternative explanation other than CAA (e.g., structural brain lesion, atrial fibrillation, extracranial, or intracranial stenosis)
mortality or dependance at 12 and 24 months | 12 and 24 months
  Mortality and dependence defined by a modified Rankin scale >2
Cognitive decline at 12 and 24 months | 12 and 24 months
  moderate or severe vascular cognitive disorders (VCD) according to the VASCOG criteria.
New MRI hemorrhagic lesion at 12 months | 12 months
  Presence of new symptomatic or asymptomatic hemorrhagic lesion (ICH, microbleeds, convexity subarachnoid hemorrhage) on follow-up MRI at 12 months
Extent of cortical superficial siderosis at 12 months | 12 months
  Extent of cSS is assessed on follow up MRI at 12 months according to the current guidelines: 0: no cSS; 1: focal cSS (restricted to ≤3 sulci); 2: disseminated cSS (≥4 sulci).
frequency of APOE ε2 and ε4 allele | baseline
  frequency of both ε2 and ε4 allele on Apolipoprotein E (APOE) genotype at baseline

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas RAPOSO, MD, Principal Investigator — University Hospital, Toulouse; Lionel CALVIERE, Principal Investigator — University Hospital, Toulouse
Locations (4):
- France (4):
  - Pellegrin Hospital, Bordeaux
  - Gui de Chauliac Hospital, Montpellier
  - Lariboisière Hospital, Paris
  - CHU Purpan. Hôpital Pierre-Paul Riquet, Toulouse

IPD SHARING:
Plan to Share IPD: No